CLINICAL TRIAL: NCT03520452
Title: Effect of Chlorogenic Acids on the Human Vasculature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 1716NRC
Record Dates: First submitted 2018-03-01; First posted 2018-05-09 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Endothelial Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- 302 mg green coffee extract (Experimental): Green coffee extract
  Interventions: Other: Green coffee extract
- 604 mg green coffee extract (Experimental): Green coffee extract
  Interventions: Other: Green coffee extract
- 906 mg green coffee extract (Experimental): Green coffee extract
  Interventions: Other: Green coffee extract

INTERVENTIONS:
Other: Green coffee extract — Reconstituted in water and given to subjects
  Arms: 302 mg green coffee extract; 604 mg green coffee extract; 906 mg green coffee extract
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study evaluates effects of different doses of chlorogenic acids on vascular health.

DETAILED DESCRIPTION:
It has been suggested that consumption of food rich in chlorogenic acids can help to improve vascular health, measured by flow mediated dilation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or postmenopausal female healthy volunteers aged 45-65 years old
2. Willing and able to sign written informed consent prior to trial entry
3. Healthy as determined by the medical history and physical examination

Exclusion Criteria:

1. Premenopausal women
2. Current smokers
3. Abnormal blood pressure, defined as follow: systolic <90 or >140 mmHg and diastolic <60 or >90 mmHg
4. Regular consumption of cholesterol-lowering medication
5. Regular consumption of antihypertensive medication
6. Regular consumption of any vasoactive medication that cannot be discontinued for at least 4 half-lives before the FMD assessment
7. Any food allergies
8. Any intakes of multivitamin-tablets and other supplemental compounds within 10 days of the study start and throughout the study
9. Inability to refrain from coffee/tea and alcohol consumption for 12 h prior to study visits
10. Acute or chronic major psychiatric illness or other major illness that in the opinion of the investigator would make the subjects' participation in the study unsafe or prevent them from fully complying with the study procedures
11. Use of medication to treat psychiatric illness (depression) within 3 months prior to the study
12. Recent significant weight loss or gain (>6% of body weight) in the past 3 months
13. Body mass index (BMI) outside 18-32 kg/m2 range
14. Alcohol intake > 280g/week (21-28 glasses per week)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Efficacy by oral administration of chlorogenic acid in improving endothelial function | 24 hours
  The primary outcome will be the average change from baseline (i.e. predose) in the %Flow Mediated Dilation

SECONDARY OUTCOMES:
Cmax of the different chlorogenic acid metabolites | 24 hours
  link for endothelial function improvement
Area Under Curve of the concentration/time curve | 24 hours
  Area Under Curve of the concentration/time curve
Tmax | 24 hours
  link for endothelial function improvement
elimination half-life. | 24 hours
  link for endothelial function improvement

OTHER OUTCOMES:
Blood concentrations in plasma. | 24 hours
  Blood concentrations in plasma.
Safety of the investigational product | from first dose till last visit
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Tan, Study Chair — Société des Produits Nestlé (SPN)
Locations (1):
- University of Western Australia, Crawley, Perth, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naylor LH, Zimmermann D, Guitard-Uldry M, Poquet L, Leveques A, Eriksen B, Bel Rhlid R, Galaffu N, D'Urzo C, De Castro A, Van Schaick E, Green DJ, Actis-Goretta L. Acute dose-response effect of coffee-derived chlorogenic acids on the human vasculature in healthy volunteers: a randomized controlled trial. Am J Clin Nutr. 2021 Feb 2;113(2):370-379. doi: 10.1093/ajcn/nqaa312. PMID 33330899